CLINICAL TRIAL: NCT05266547
Title: Impact of Optical Coherence Tomography on Long-term Clincal Outcomes in Patients With Acute Myocardial Infarction
Brief Title: Impact of OCT on Outcomes in AMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Luhe Hospital (Other)
Responsible Party: Principal Investigator, Jincheng Guo, chairman of CCU, Beijing Luhe Hospital
Other Study IDs: BeijngLH
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Acute Myocardial Infarction
Keywords: Tomography, Optical Coherence; STEMI; NSTEMI; Major adverse cardiovascular event
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OCT guided group
  Interventions: Device: OCT guided coronary intervention
- angiography guided group
  Interventions: Device: OCT guided coronary intervention

INTERVENTIONS:
Device: OCT guided coronary intervention — patients were divided into two groups,on OCT guided coronary group and coronary angiography guided group

SUMMARY:
This protocol describes a retrospective, single-center study intended to test the impact of optical coherence tomography(OCT) on long term clincical outcomes in patients with acute myocardial infarction(AMI). All the patients will be followed by intracoronary OCT at medium follow-up of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old
* Patients undergo cardiac catheterization and percutaneous coronary intervention(PCI) for AMI(STEMI or NSTEMI) ST-segment elevation myocardial infarction was defined according to the universal definition of myocardial infarction, symptoms onset≤ 24h.NSTEMI was defined as elevated troponin levels and the absence of ST elevation at the time of diagnosis, PCI was performed within 24hours after symtoms onset.
* Sufficient quality of the OCT recording allowing for CoreLab analysis.

Exclusion Criteria:

* ostial of Left main disease
* Cardiogenic shock or severe hemodynamic instability
* Severe renal insufficiency (creatinine clearance ≤30 mL/min)
* Bacteraemia or septicaemia
* Severe coagulation disorders
* Patients with life expectancy less than 1 year
* Patients who refuse to sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this retrospective study, all the patients ≥18yesrs with AMI enrolled was devided into 2 groups, the primary endpoint will be major adverse cardiovascular events at least 3 years clinical follow up.
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiovascular event | 3 year
  including cardiovascualr death, myocardial infarction, and target lesion revascularization, target vessel revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Luhe Hospital, Beijing, China